CLINICAL TRIAL: NCT00308152
Title: Randomised, Controlled Trial of Intravenous Saline Pre-hydration in Patients Undergoing Outpatient Colonoscopy
Brief Title: Intravenous Saline Pre-hydration in Patients Undergoing Outpatient Colonoscopy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Canberra Hospital (Other)
Responsible Party: Principal Investigator, Dr Douglas Taupin, Senior Staff Specialist, The Canberra Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 11/05.851
Record Dates: First submitted 2006-03-28; First posted 2006-03-29 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Colonic Diseases
Keywords: Colonoscopy; Rehydration; Sedation
MeSH Terms: conditions — Colonic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Observation only
- Active (Active Comparator): Infusion of 1 liter normal saline before sedated colonoscopy
  Interventions: Drug: Infusion of 1 litre of normal saline before colonoscopy

INTERVENTIONS:
Drug: Infusion of 1 litre of normal saline before colonoscopy — Prehydration with normal saline
  Arms: Active

SUMMARY:
Colonoscopy and sedation are frequently accompanied by hypotension, which reduces the amount of sedation able to be employed. Blood pressure is restored by the infusion of intravenous normal saline. Prophylactic infusion of normal saline may enhance the colonoscopy completion rate, and patient comfort during colonoscopy and during the recovery from colonoscopy.

The investigators propose randomising consenting adult patients attending outpatient colonoscopy to one of two treatment arms:

(i) A control arm

(ii) A treatment arm, with pre-hydration with an infusion of 1.0 litre of normal saline immediately prior to colonoscopy.

Outcome measures include colonoscopy completion rates, hypotension during or after colonoscopy, and patient ratings of comfort and satisfaction.

DETAILED DESCRIPTION:
Outpatient colonoscopy is a generally well-tolerated elective procedure. Colonoscopy completion rate is governed in part by patient comfort, which is enhanced by adequate sedation. In addition, comfort following colonoscopy determines timely recovery from the procedure and return to usual activities.

Colonoscopy and sedation are frequently accompanied by hypotension (systolic blood pressure less than 100 mm Hg), which reduces the amount of sedation able to be employed. Where apparent, blood pressure is restored by infusion of intravenous normal saline. We have observed that hypotension is relatively common and may be present at or shortly after the commencement of the procedure, suggesting that many patients undergoing colonoscopy have reduced blood volume. Therefore, prophylactic infusion of normal saline may enhance colonoscopy completion rate, and patient comfort during colonoscopy and during recovery from colonoscopy.

We propose randomising consenting adult patients attending outpatient colonoscopy to one of two treatment arms:

(i) A control arm, with standard sedation and monitoring during colonoscopy, and infusion of normal saline if systolic BP ≤ 95 mmHg for more than 3 minutes (two observation periods) until completion of the procedure;

(ii) A treatment arm, with pre-hydration with an infusion of 1.0 litre of normal saline immediately prior to colonoscopy.

Outcome measures include colonoscopy completion rates, hypotension during or after colonoscopy, and patient ratings of comfort and satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or older
* Able to provide informed consent
* Booked for outpatient colonoscopy, where appointment has been generated by Gastroenterology Unit bookings staff.

Exclusion Criteria:

* Booked for anaesthetist-supervised colonoscopy because of previous sedation difficulties or significant co-morbidity (American Society of Anesthesiology Class III or IV)
* Subjects requiring dialysis
* Subjects receiving parenteral nutrition
* Subjects with current congestive cardiac failure
* Subjects with conditions preventing placement and accurate use of the automatic blood pressure cuff on the left arm, such as morbid obesity or lymphoedema

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2006-02; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
The number of subjects with documented hypotension (systolic blood pressure [BP] ≤ 95 mmHg for 1 or more automatic BP measures taken at 3 minute intervals), during colonoscopy or the recovery period
Colonoscopy completion rates. Raw completion rates, with no allowance for failed bowel preparation or technical difficulties, will be used.
The number of subjects reaching criteria for discharge at 30 minutes after arrival in the recovery area
Comfort and satisfaction scores: discomfort during colonoscopy, discomfort after colonoscopy, satisfaction with sedation, overall satisfaction
Time taken to resume normal activities
Where relevant, adverse events such as post-procedure nausea, syncope, and prolonged recovery time, will be recorded in both arms of the study for comparison.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas R Taupin, MBBS, PhD, Principal Investigator — The Canberra Hospital
Locations (1):
- The Canberra Hospital, Garran, Australian Capital Territory, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rex DK, Heuss LT, Walker JA, Qi R. Trained registered nurses/endoscopy teams can administer propofol safely for endoscopy. Gastroenterology. 2005 Nov;129(5):1384-91. doi: 10.1053/j.gastro.2005.08.014. PMID 16285939
- [Background] Heuss LT, Schnieper P, Drewe J, Pflimlin E, Beglinger C. Risk stratification and safe administration of propofol by registered nurses supervised by the gastroenterologist: a prospective observational study of more than 2000 cases. Gastrointest Endosc. 2003 May;57(6):664-71. doi: 10.1067/mge.2003.191. PMID 12709694
- [Background] Schrier RW. Body fluid volume regulation in health and disease: a unifying hypothesis. Ann Intern Med. 1990 Jul 15;113(2):155-9. doi: 10.7326/0003-4819-113-2-155. PMID 2193561
- [Background] Ristikankare M, Julkunen R, Laitinen T, Wang SX, Heikkinen M, Janatuinen E, Hartikainen J. Effect of conscious sedation on cardiac autonomic regulation during colonoscopy. Scand J Gastroenterol. 2000 Sep;35(9):990-6. doi: 10.1080/003655200750023093. PMID 11063163
- [Background] Chen SC, Rex DK. Review article: registered nurse-administered propofol sedation for endoscopy. Aliment Pharmacol Ther. 2004 Jan 15;19(2):147-55. doi: 10.1111/j.0269-2813.2004.01833.x. PMID 14723606
- [Background] Sipe BW, Rex DK, Latinovich D, Overley C, Kinser K, Bratcher L, Kareken D. Propofol versus midazolam/meperidine for outpatient colonoscopy: administration by nurses supervised by endoscopists. Gastrointest Endosc. 2002 Jun;55(7):815-25. doi: 10.1067/mge.2002.124636. PMID 12024134